CLINICAL TRIAL: NCT00449358
Title: Correlation Between Mohs Surgery and Microscopic Fluorescence Photometry in Determination of Histological Borders in Basal Cell Carcinoma .
Brief Title: Checking Wether the m-ALA Cream Could Mark Correctly the Borders of BCC's Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assuta Hospital Systems (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2006-01

CONDITIONS: Basal Cell Carcinoma
Keywords: bcc
MeSH Terms: conditions — Carcinoma, Basal Cell

INTERVENTIONS:
Procedure: apply methyl-ALA cream

SUMMARY:
Correlation between Mohs surgery and microscopic fluorescence photometry in determination of histological borders in Basal Cell Carcinoma .

DETAILED DESCRIPTION:
Background: Basal Cell Carcinoma (BCC) is the most common form of nonmelanoma skin cancer worldwide. BCCs are slow-growing, locally invasive tumors that rarely metastasize but can cause extensive morbidity through local tissue destruction. Recurrence is often the consequence of incomplete removal of the cancer tissue. Mohs' micrographic surgery is considered the most effective treatment modality for BCC with a recurrence rate of less than 5 %, however, the technique requires specialized training and is labor-intensive and costly. Fluorescence imaging by topical application of a tumor-localizing agent such as methyl 5-aminolevulinic acid (MAL), resulting in buildup of photosensitizing porphyrin IX (PpIX) that can be visualized by Woods' light fluorescence, might serve as a quick and simple "bed-side" technique for demarcation of BCC tumor borders prior to surgical excision Objective: To test the reliability of MAL-induced porphyrin fluorescence tumor demarcation by comparison with the tumor borders determined by Mohs' surgery Methods: Twenty eight patients with facial BCCs (17 nodular, 3 superficial, 1 morphea type, 3 ulcerated and 4 recurrent tumors) scheduled for Mohs' surgery were recruited for the study. The night before the surgical procedure, crusts were gently removed and an approximately 1 mm thick layer of a cream containing 16 % MAL (MetvixR) was applied to the tumor area as well as to the surrounding skin and covered by a transparent occlusive dressing. The following morning (10-17 hours after MetvixR application), the dressing was removed, and the lesion size was determined with a caliber by measuring the largest perpendicular diameters under natural (clinical size) and Woods' (fluorescence size) illumination. The patients then underwent the scheduled Mohs' surgical procedure, and the tumor size (Mohs' size) was determined when reaching the tumor free margins.

ELIGIBILITY:
Inclusion Criteria:

* A- bove 18 years

Exclusion Criteria:

* Childern
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-02; Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
comparing the tumor area measured with the PDD thechnique and the actual tumor size found at the end of the Mohs surgery

CONTACTS AND LOCATIONS:
Overall Officials: Enk David, m.d, phd, Principal Investigator — Hadassah ein-karem university hospital
Locations (1):
- Assuta hospital, Tel Aviv, Israel